CLINICAL TRIAL: NCT06962072
Title: Body Image, Health-related Quality of Life, and Function After Soft Tissue Sarcoma Resection
Brief Title: Outcomes Following Limb Sparing Surgery for Soft Tissue Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Floortje Verspoor, Clinical researcher, Amsterdam UMC, location AMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL85908.018.23
Record Dates: First submitted 2025-03-28; First posted 2025-05-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Body image; Quality of life; Function; Functioning
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivors following the resection of extremity soft tissue sarcoma: Patients who were treated with surgical resection for primary non-metastatic extremity STS at the Amsterdam UMC between 2010 and 2021.
  Interventions: Procedure: Surgical resection with or without radiotherapy and/or chemotherapy

INTERVENTIONS:
Procedure: Surgical resection with or without radiotherapy and/or chemotherapy — The surgical resection of STS serves as the primary treatment, aiming to completely remove the tumor with a wide margin of surrounding healthy tissue to minimize the risk of recurrence. Radiotherapy and/or chemotherapy may be incorporated depending on the tumor's type, stage, and grade.

SUMMARY:
The goal of this study is to assess body image, health-related quality of life (QoL), and functioning (gait function, joint function, and walking ability) in patients after resection of localized soft tissue sarcoma (STS) of the extremities. A secondary objective is to assess the influence of different variables (e.g., radiotherapy, ethnicity, etc.) on body image, health-related QoL, and functioning.

Patients who underwent a surgical resection at the Amsterdam UMC between 2010 and 2021 will be approached to participate in the study. Participants will complete four questionnaires and undergo a physical examination. Additionally, they will have a 3D gait analysis, a 6-minute walk test with gas analysis, and a muscle strength assessment. Furthermore, muscle volume change will be evaluated on pre- versus postoperative MRI scans.

DETAILED DESCRIPTION:
Primary objectives :

* To assess body image, health-related QoL, self-reported activity limitations, and pain after STS resections as defined in the The International Classification of Functioning, Disability and Health (ICF) domains.
* To assess the functioning of the patients after STS resections as defined by the ICF domains of body function, body structure, and activities and participation:
* Body function:

  1. Evaluate impairments in gait biomechanics.
  2. Evaluate impairments in joint function as determined by range of motion and muscle strength.
* Body structure:

  a. Evaluate muscle volume change on pre- and postoperative MRI scans and correlate these findings with body image, health-related quality of life, activity limitations, and functional impairments.
* Activities and participation:

  1. Objectify activity limitations by walking speed, and energy cost.
  2. Objectify balance and mobility as measured by Timed Up and Go (TUG) test and Timed Up and Down Stairs (TUDS) test.

Secondary objectives:

* To identify factors associated with body image, health-related QoL and functioning in extremity STS survivors.
* To compare body image, health-related QoL and functioning between patients who were treated with and without radiotherapy.

Srudy design:

This is a cross-sectional follow-up study. All records of consecutive non-metastatic extremity STS patients who underwent surgical resection between 2010 and 2021 at the Amsterdam UMC will be evaluated. Both deceased patients and survivors are included to obtain a realistic picture of the entire population. Survivors (approximately N = 125-150) will be approached to take part in this study by phone, followed by a letter explaining the study, including an informed consent form.

At baseline, patient demographics, tumor characteristics, diagnostics, and treatments will be collected. The participants can either fill out the self-reported questionnaires at home through the internet (using EPIC/Castor) or on a tablet at the outpatient clinic with the help of the investigator.

Participants will be invited to visit the outpatient clinic for a physical examination, which will include assessments of joint range of motion, limb circumference, balance, and mobility. Balance and mobility will be evaluated using the Timed Up and Go (TUG) test and the Timed Up and Down Stairs (TUDS) test. Muscle strength will be assessed using a hand-held dynamometer and the Medical Research Council (MRC) scale. Participants can complete the computer-based questionnaires at the outpatient clinic if not already completed at home. This part of the study will take place at the Department of Orthopedic Surgery and Sports Medicine.

Additionally, participants will undergo a 3D gait analysis to assess gait biomechanics, a muscle strength assessment using a Biodex dynamometer, and a 6-minute walk test to evaluate walking speed and energy cost. These assessments will be conducted at the Department of Rehabilitation.

Depending on the test, results will be compared as follows:

* Against general population means
* Between patients who have undergone upper and lower extremity STS resection
* Between the affected limb and the contralateral healthy limb

Additionally, the results from the objective functional tests and the MRI-scans (with tumor and pre- plus postoperative muscle specific features) will be correlated with body image and health-related QoL questionnaires. To identify factors associated with body image, health-related QoL, and functioning, we will assess whether the collected factors (baseline patients and tumor characteristics, treatments, and complications) are associated with better or worse outcomes of the questionnaires and the functional tests.

ELIGIBILITY:
Inclusion Criteria:

* Treated with surgical resection for primary non-metastatic extremity STS at the Amsterdam UMC between 2010-2021.
* Being able to visit the Amsterdam UMC, location AMC once or twice.
* Pregnant patients must agree to be scheduled 5 months after their pregnancy ends.

Exclusion Criteria:

* Patients who cannot maintain 6 minutes of walking will be excluded from the 6-minute walk test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for primary non-metastatic extremity STS through surgical resection, with or without (neo-) adjuvant radiotherapy, between 2010-2021.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Gait biomechanics | Baseline
  A 3D gait analysis will be conducted. Ground reaction forces will be captured using two force plates embedded in the center of the walkway. Three valid gait trials will be collected (meaning a clear strike on the force plate(s)). For each trial, data on joint angles and net joint moments (via inverse dynamics) and powers around the hip, knee, and ankle will be calculated. Data will be averaged over three trials to represent the outcome. Also, spatiotemporal gait parameters, such as step length (m) step width (m) and walking speed (m/s} will be calculated.
Range of motion in degrees | Baseline
  Rang of motion in degrees wil be assessed during the physical examination using a goniometer
Limb circumference in cm | Baseline
  Limb circumference in cm will be measured during the physical examination
Muscle strength in newton measured with a handheld dynamometer | Baseline
  A handheld dynamometer will be used to measure muscle strength during the physical examination. The participant will be asked to lie or to sit in a specific position and resistance will be applied depending on the muscle group to be tested. The dynamometer will be held perpendicular to the tested limb and the participant will be asked to actively perform a maximum contraction against the dynamometer. The participants will be instructed to push as hard as they can, and the examiner will apply equal force to that of the participant. On each muscle group, three trials will be performed, and the highest record among the three trials will be recorded. Newton (N) will be used to express muscle strength.
Muscle strength tested with the MRC scale | Baseline
  Based on the clinician's assessment of the normal strength of the muscle group under examination, the scale rates muscle strength on a scale of 0 to 5, with 0 representing no visible contraction and 5 representing a movement against complete resistance.
Muscle strength in newton meters measured with a Biodex dynamometer. | Baseline
  Quantitative force of muscles in arms or legs will be assessed using a Biodex dynamometer. The measures will be performed on both sides. On each muscle group, three trials will be performed, and the highest recorded value will be used for the analysis. Peak torque will be calculated and recorded in newton meters (Nm). Peak torque is defined as the highest torque output produced by muscle contraction during a repetition.
Change in muscle volume between preoperative and postoperative MRI scans | Baseline
  The change in muscle volume between preoperative and postoperative MRI scans will be determined.
Walking energy cost in J/kg/m | Baseline
  Walking energy cost in J/kg/m will be determined during a 6-minute walk test with simultaneous gas analysis. The oxygen uptake (VO2) and carbon dioxide production (VCO2) are measured breath-by-breath using a portable gas analysis system. First, the energy consumption will be measured for 8 minutes while the subjects are sitting on a chair. Then, the energy cost will be measured while subjects are walking during a 6-minute walk test at a comfortable, self-selected speed on an indoor oval route.
Walking speed in m/s | Baseline
  Walking speed wil be assessed during the 6-minute walk test. It will be measured and calculated as the average speed over the steady state period.
Time Up and Go (TUG) test | Baseline
  In the TUG test, the time (in seconds) required for a patient to get up from a chair, walk 3 meters to a marked point on the ground, turn, walk back to the chair, and sit down will be recorded.
Timed Up and Down Stairs (TUDS) test | Baseline
  In the TUDS test, the time (in seconds) required for a patient to go up a flight of stairs quickly and safely, turn around on the top step, and descend to the bottom step with both feet landing on the ground will be recorded.
Body image as assessed by the Body Image Scale (BIS) | Baseline
  Body image after STS resection will be evaluated with the Body Image Scale (BIS). This questionnaire consists of 10 questions about body image. For each question, the patient has to choose between 'not at all' (score 0), 'a little' (score 1), 'quite a bit' (score 2), and 'very much' (Score 3). In total, a score between 0 and 30 can be achieved with 0 indicating no distress or symptoms and 30 indicating the highest level of distress and symptoms
Health-related quality of life (QoL) as assessed by the Patient Reported Outcome Measurement Information System-Computerized Adaptive Test (PROMIS-CAT) | Baseline
  Health-related QoL and activity limitations will be assessed using the PROMIS-CAT health domains: physical functioning, social role participation, pain interference, fatigue, upper extremity, and emotional distress (anxiety and depression). PROMIS instruments are scored with T-scores, which are standardized to the general population. The average of the reference population is set at 50 points, with a standard deviation of 10.
Quality of life as assessed by the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) questionnaire | Baseline
  This questionnaire is divided into two sections: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system consists of five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are five levels for each dimension. Patients will be asked to check the box next to the most suitable statement in every one of the five dimensions. For the EQ-VAS, patients will assess their health on a vertical visual analogue scale from 0 to 100 (0 being the worst and 100 being the best imaginable health).
Level of pain as assessed by the Numeric Rating Scale (NRS) | Baseline
  The level of pain will be assessed using the Numeric Rating Scale (NRS) 0 to 10. The pain will be measured at four intervals, with 0 being no pain at all and 10 being the worst pain imaginable: currently (1), average last week (2), severity pain when worst (3) or least (4).

SECONDARY OUTCOMES:
Patient demographics | Baseline
  At baseline patiënt demographics (e.g age, sex, marital status, educational level, occupational status, ethnicity, country of origin and smoking status) will be collected
Body Mass Index (BMI) in kg/m2 | Baseline
  BMI in kg/m² will be calculated as weight (kg) divided by height squared (m²)
Tumor characteristics | Baseline
  At baseline, tumor characteristics (e.g. tumor subtype, grade, stage and location) will be collected.
Tumor size in cm | Baseline
  Tumor size in cm will be measured on the pre-operative MRI scan
Tumor volume in cm³ | Baseline
  Tumor volume in cm³ will be measured on the pre-operative MRI scan
Involvement of adjacent structures | Baseline
  Tumor invasion of adjacent stucrures will be assessed on the pre-operative MRI scan.
Tumor depth | Baseline
  Tumor depth (deep or superficial) will be assessed on the pre-operative MRI scan.
Treatments | Baseline
  At baseline, data on treatments (surgery, radiotherapy, and chemotherapy) will be recorded
Complications | Baseline
  Treatment-related complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD will not be made pubicly available but can be obtained upon request at the study's sponsor. When a valid reason for the re-use of study data is provided, a Data Sharing Agreement can be set up.